CLINICAL TRIAL: NCT03653429
Title: Efficacy of Tranexamic Acid in Foot and Ankle Surgeries- a Randomized Controlled Trial.
Brief Title: Efficacy of Tranexamic Acid in Foot and Ankle Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Yan Lai, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 17-1691
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Results first posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Foot and Ankle Surgeries; Bunion
Keywords: foot and ankle surgeries; tranexamic acid; wound healing; blood loss
MeSH Terms: conditions — Bunion; Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid group (Active Comparator): 10mg/kg intravenous tranexamic
  Interventions: Drug: Tranexamic Acid
- Normal Saline group (Placebo Comparator): 10mg/kg intravenous normal saline
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Tranexamic Acid — administered prior to surgical incision
  Arms: Tranexamic acid group
Drug: Normal saline — administered prior to surgical incision
  Arms: Normal Saline group

SUMMARY:
Epidemiology of foot and ankle surgeries that present to the hospitals in the US are often underestimated. However there has been growing emphasis on identification of these injuries and practice patterns.

DETAILED DESCRIPTION:
Approximately 20% of all foot and ankle fractures are open. Excellent operative field without measurable bleeding remain prerequisite of most orthopedic procedures. Increase blood loss can increase the risk of infection, hematoma formation and wound complications. Presence of blood in synovium not only has direct corrosive effects but also causes increased intra capsular pressure leading to capsular fibrosis culminating as ankyloses.

Tourniquets are employed to optimize surgical field visualization thereby limiting operative duration and improving technical precision. There are several unwanted effects that can arise from use of tourniquet like neurapraxia, vascular injury, post operative swelling etc. Hence there is a growing interest in achieving the same operative goals without the use of tourniquet.

Antifibrinolytics come to one's rescue to achieve a blood sparing effect. Its efficacy in reducing intra operative and post operative blood loss is well documented in cardiac surgery, hip and knee replacement surgery and spinal surgery. Tranexamic acid is a synthetic antifibrinolytic drug that competitively blocks the lysine-binding sites of plasminogen, plasmin and tissue plasminogen activator, thereby delaying fibrinolysis and blood clot degradation. It has been effectively used as IV, oral, topical as well as intra articular dosing. The effects of IV administration lasts 8-17 hours after the initial dose. Orthopedic surgeons have incorporated TXA into multiple elective surgeries as a means of reducing blood loss and transfusion requirements. Reduced bleeding translates to decreased incidence of wound hematoma and other complications.

Effectiveness of Tranexamic acid(TXA) is unknown in foot and ankle surgeries. The aim of this study is to not only evaluate effectiveness of intravenous TXA in reducing post operative blood loss during foot and ankle surgeries but also if it modulates to reduced wound complications and reduced narcotic consumption.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiology) class I-IV
* age 8-75.

Exclusion Criteria:

* ASA class V
* morbid obesity
* patient refusal
* patients with known coagulopathy disorder
* renal insufficiency
* hepatic dysfunction
* serious cardiac disease
* an allergy to TXA or receiving antiplatelet and /or anticoagulant drugs will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ettore Vulcano, MD, Principal Investigator — Ichan School of Medicine
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Ichan School of Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xie B, Tian J, Zhou DP. Administration of Tranexamic Acid Reduces Postoperative Blood Loss in Calcaneal Fractures: A Randomized Controlled Trial. J Foot Ankle Surg. 2015 Nov-Dec;54(6):1106-10. doi: 10.1053/j.jfas.2015.07.006. Epub 2015 Aug 24. PMID 26310621

RESULTS

PARTICIPANT FLOW:
Groups:
- Tranexamic Acid Group: 10mg/kg intravenous tranexamic acid administered prior to surgical incision
- Normal Saline Group: 10mg/kg intravenous normal saline administered prior to surgical incision
Period: Overall Study
Arm/Group | Tranexamic Acid Group | Normal Saline Group
Started | 49 | 51
Completed | 45 | 41
Not Completed | 4 | 10
Not completed — Physician Decision | 4 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid Group | Normal Saline Group | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.24 (15.49) | 52.51 (14.05) | 51.89 (14.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 18 | 18 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 37 | 39 | 76
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Estimated Blood Loss
Description: Total estimated blood loss in millilitres during the surgery
Time Frame: Average intra operative time 1-2 hours
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Tranexamic Acid Group | Normal Saline Group
Number analyzed (Participants) | 49 | 51
ml | 40.41 (136.78) | 18.75 (49.40)

2. Secondary Outcome: Number of Participants With Wound Complications
Description: Number of participants with wound complications at first post-operative visit and at 2 weeks post surgery
Time Frame: at first post-operative visit, 2 weeks post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Group | Normal Saline Group
Number analyzed (Participants) | 49 | 51
Participants
  first post-operative visit | 8 | 8
  2 weeks post surgery | 8 | 8

3. Secondary Outcome: Intra Operative Narcotic Consumption
Description: Total intraoperative narcotic consumption in terms of morphine equivalents.(mme)
Time Frame: Average intra operative time 1-2 hours
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Tranexamic Acid Group | Normal Saline Group
Number analyzed (Participants) | 49 | 51
MME | 93.37 (58.80) | 125.40 (79.17)

4. Secondary Outcome: Post Operative Narcotic Consumption
Description: Post operative narcotic consumption, morphine mili equivalents
Time Frame: 2 weeks after surgery
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Tranexamic Acid Group | Normal Saline Group
Number analyzed (Participants) | 49 | 51
MME | 6.12 (13.32) | 10.10 (22.21)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Tranexamic Acid Group | Normal Saline Group
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 0/49 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT03653429/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT03653429/ICF_001.pdf